CLINICAL TRIAL: NCT01584362
Title: Phase I Study of Oxfendazole (Toward the Treatment of Neurocysticercosis)
Brief Title: Single Ascending Dose Safety Study of Oxfendazole
Acronym: OXFEND-02
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study conducted under Clinical Trials Agreement as NIAID registration NCT02234570
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); School of Veterinary Medicine, Universidad Nacional Mayor de San Marcos (Unknown)
Responsible Party: Principal Investigator, Robert Gilman, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXFEND-02, IND 113,628; IND 113,628 (Other: FDA)
Record Dates: First submitted 2012-04-18; First posted 2012-04-25 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Tenia Solium Infection
Keywords: Taenia solium; neurocysticercosis; oxfendazole; clinical trial, phase 1; safety; pharmacokinetics
MeSH Terms: conditions — Taeniasis; Neurocysticercosis | interventions — oxfendazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- oxfendazole 0.3 (Experimental): administration of a single oral 0.3mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole
- placebo comparator (Placebo Comparator): administration of a single oral dose of placebo
  Interventions: Drug: placebo
- oxfendazole 1.0 (Experimental): administration of a single oral 1.0 mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole
- oxfendazole 3.0 (Experimental): administration of a single oral 3 mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole
- oxfendazole 10 (Experimental): administration of a single oral 10 mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole
- oxfendazole 20 (Experimental): administration of a single oral 20 mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole
- oxfendazole 30 (Experimental): administration of a single oral 30 mg/kg dose of oxfendazole
  Interventions: Drug: oxfendazole

INTERVENTIONS:
Drug: oxfendazole — administration of a single oral 1.0 mg/kg dose of oxfendazole
  Arms: oxfendazole 1.0
Drug: placebo — single oral dose of placebo
  Arms: placebo comparator
Drug: oxfendazole — administration of a single oral 3.0 mg/kg dose of oxfendazole
  Arms: oxfendazole 3.0
Drug: oxfendazole — administration of a single oral 0.3 mg/kg dose of oxfendazole
  Arms: oxfendazole 0.3
Drug: oxfendazole — administration of a single oral 10 mg/kg dose of oxfendazole
  Arms: oxfendazole 10
Drug: oxfendazole — administration of a single oral 20 mg/kg dose of oxfendazole
  Arms: oxfendazole 20
Drug: oxfendazole — administration of a single oral 30 mg/kg dose of oxfendazole
  Arms: oxfendazole 30

SUMMARY:
This research is being done to learn about the safety in humans of a medicine that is already used in cows and pigs to treat worms. The medicine may be useful for people who have these or other worms. The medicine will be studied first in healthy people, who will be given a very small amount of the medicine once. If the smallest amount of medicine is found to be safe, a slightly higher amount will be given to a new group of volunteers. The highest amount that will be tested is similar to the amount given to animals. If the medicine can be given safely to healthy people in the planned amounts, a later study will be done in people who have worms to see if the medicine kills the worms.

DETAILED DESCRIPTION:
The Phase I study proposed is a randomized, double-blind, placebo-controlled evaluation of the safety and pharmacokinetics of escalating single oral doses of oxfendazole (0.3 to 30 mg/kg) in healthy volunteers. The dose will be increased approximately three-fold (one-half log) at each increment, and each cohort will comprise ten volunteers (eight drug, two placebo). Subjects will be monitored for three weeks after dosing, including monitoring the pharmacokinetics and metabolism of oxfendazole in blood and urine. Each new cohort will be dosed only after the three week safety data for the preceding group have been analyzed. If a clinically significant adverse event is observed, and if this event is possibly drug-related, an additional (and final) cohort of volunteers will repeat the highest tolerated dose of oxfendazole. Up to 70 volunteers (56 drug, 14 placebo) will complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Height and weight within 25% of means for his/her gender and age.
* Willing to use two acceptable methods of contraception (approved oral, injectable, or implantable drug, IUD, diaphragm or condom with spermicidal jelly or foam, or sexual abstinence) for a minimum of one week before, and three weeks after dosing with oxfendazole; or surgically sterile.
* Able to give written informed consent.
* Able to provide a home phone number, and the name, address, and phone number of a person willing to assist making contact during the follow-up phase of the study.

Exclusion Criteria:

* Pregnant.
* Breast feeding.
* Chronic drug/alcohol user.
* Has clinically significant abnormalities in screening examinations
* Has history of sensitivity to related benzimidazole compounds (e.g. albendazole, mebendazole).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
serious adverse events | up to three weeks after dosing
  Proportion of patients who present with serious adverse events (SAEs) related to oxfendazole.

SECONDARY OUTCOMES:
adverse events | up to three weeks after dosing
  proportion of subjects who present with adverse events (AEs) related to ocfendazole
Pharmacokinetic Profile | blood samples are drawn at 17 time points up to three weeks and urine is collected at 7 intervals up to 72 hours after dosing
  The following PK parameters will be analyzed:
  Maximum plasma concentration (Cmax), Time to Cmax (Tmax), Elimination rate constant (Iz), Elimination half-life (T½), Area under the curve to the final sample (AUC0-t), Area under the curve to infinity (AUC∞), Oral clearance (CL/F), Oral volume of distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Gilman, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Result] Gonzalez AE, Falcon N, Gavidia C, Garcia HH, Tsang VC, Bernal T, Romero M, Gilman RH. Treatment of porcine cysticercosis with oxfendazole: a dose-response trial. Vet Rec. 1997 Oct 18;141(16):420-2. doi: 10.1136/vr.141.16.420. PMID 9364715
- [Result] Gonzales AE, Garcia HH, Gilman RH, Gavidia CM, Tsang VC, Bernal T, Falcon N, Romero M, Lopez-Urbina MT. Effective, single-dose treatment or porcine cysticercosis with oxfendazole. Am J Trop Med Hyg. 1996 Apr;54(4):391-4. doi: 10.4269/ajtmh.1996.54.391. PMID 8615453
- [Result] Gonzalez AE, Falcon N, Gavidia C, Garcia HH, Tsang VC, Bernal T, Romero M, Gilman RH. Time-response curve of oxfendazole in the treatment of swine cysticercosis. Am J Trop Med Hyg. 1998 Nov;59(5):832-6. doi: 10.4269/ajtmh.1998.59.832. PMID 9840607